CLINICAL TRIAL: NCT03168295
Title: SGLT2 INHIBITION AND STIMULATIION OF ENDOGENOUS GLUCOSE PRODUCTION Significance - PROTOCOL 3: Role of the Renal Nerves in the Increase in EGP in Response to Glucosuria
Brief Title: PROTOCOL 3: Role of the Renal Nerves in the Increase in EGP in Response to Glucosuria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HSC20160042H; R01DK107680 (NIH)
Record Dates: First submitted 2017-05-24; First posted 2017-05-30 (Actual); Results first posted 2020-01-14 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Post renal transplant type 2 diabetes mellitus patients and non-diabetic mellitus patients after renal transplant with a control group of type 2 diabetes mellitus who have not undergone renal transplant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo first and then dapagliflozin (Experimental): Renal transplant subjects with intact native kidneys with Type 2 Diabetes Mellitus receive dapagliflozin then placebo
  Interventions: Drug: Dapagliflozin 10mg then Placebo Oral Tablet; Drug: Placebo Oral Tablet then Dapagliflozin 10mg
- Dapagliflozin first then placebo (Active Comparator): Renal transplant subjects with intact native kidneys who are non-diabetic receive placebo then dapagliflozin
  Interventions: Drug: Dapagliflozin 10mg then Placebo Oral Tablet; Drug: Placebo Oral Tablet then Dapagliflozin 10mg
- Control Group (Other): Subjects who are type 2 diabetes mellitus who have not undergone renal transplant.
  Interventions: Drug: Dapagliflozin 10mg then Placebo Oral Tablet

INTERVENTIONS:
Drug: Dapagliflozin 10mg then Placebo Oral Tablet — SGLT2 inhibitor - Dapagliflozin then Placebo
  Other Names: Farxiga then placebo
Drug: Placebo Oral Tablet then Dapagliflozin 10mg — Placebo then SGLT2 inhibitor - Dapagliflozin
  Other Names: Placebo then Farxiga
  Arms: Dapagliflozin first then placebo; Placebo first and then dapagliflozin

SUMMARY:
Purpose/Objectives: Examining the effect of SGLT2 inhibition on EGP and plasma glucose concentration in diabetic and non-diabetic subjects after kidney transplantation (i.e. renal denervation) or in subjects after renal sympathectomy (63) can add insight about the possible role of a neural arc which mediates the changes in plasma glucagon and/or insulin concentration in response to glucosuria.

DETAILED DESCRIPTION:
Purpose/Objectives: Examining the effect of SGLT2 inhibition on EGP and plasma glucose concentration in diabetic and non-diabetic subjects after kidney transplantation (i.e. renal denervation) or in subjects after renal sympathectomy (63) can add insight about the possible role of a neural arc which mediates the changes in plasma glucagon and/or insulin concentration in response to glucosuria.

Research Design/Plan: After screening, eligible subjects will receive 2 measurements of endogenous glucose production with a prime-continuous infusion of 3-3H-glucose. Each measurement will be performed on a separate day in random order after a 10-12 hour overnight fast and will last 8 hours (from 6 AM to 2 PM). After a 3-hour tracer equilibration period, each subject will receive one of the following medications in random order: (i) placebo and (ii) dapagliflozin 10 mg. Following the test medication at 9 AM, blood samples will be drawn every 20 minutes for an additional 5 hours and plasma glucose, insulin, C-peptide, glucagon, catecholamine concentrations and tritiated glucose sp act will be measured.

Methods: Visit 1: Screening Visit 2: Endogenous Glucose Production Measurement (EGP) Visit 3: After completing the first EGP measurement, subjects will return to the Diabetes Research Unit for the second study.

ELIGIBILITY:
Inclusion Criteria:

* age = 18-70 years
* BMI = 18.5-40 kg/m2
* HbA1c ≥ 7.0% and ≤10.0% for type 2 diabetics
* males or females
* Must be at least 3 months post renal transplantation and be on a stable dose of prednisone (≤5 mg/day), tacrolimus, and mycophenolate mofetil
* Not taking any antidiabetic medications or who are treated with metformin, sulfonylurea, dipeptidyl peptidase 4 (DPP4) inhibitor, thiazolidinedione or some combination
* Must be in good general health as determined by physical exam, medical history, blood chemistries, CBC, TSH, T4, EKG and urinanalysis

Exclusion Criteria:

* Subjects who are taking insulin or SGLT2 inhibitor are excluded
* Only subjects whose body weight has not been stable (± 3 lbs) over the preceding three months and/or who participate in an excessively heavy exercise program will be excluded.
* Individuals with evidence of proliferative diabetic retinopathy, plasma creatinine >1.4 females or >1.5 males (and eGFR <45ml/min.1.73m2), or 24-hour urine albumin excretion > 300 mg will be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph A DeFronzo, MD, Principal Investigator — The University of Texas Health Science at San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daniele G, Solis-Herrera C, Dardano A, Mari A, Tura A, Giusti L, Kurumthodathu JJ, Campi B, Saba A, Bianchi AM, Tregnaghi C, Egidi MF, Abdul-Ghani M, DeFronzo R, Del Prato S. Increase in endogenous glucose production with SGLT2 inhibition is attenuated in individuals who underwent kidney transplantation and bilateral native nephrectomy. Diabetologia. 2020 Nov;63(11):2423-2433. doi: 10.1007/s00125-020-05254-w. Epub 2020 Aug 22. PMID 32827269
- [Derived] Solis-Herrera C, Daniele G, Alatrach M, Agyin C, Triplitt C, Adams J, Patel R, Gastaldelli A, Honka H, Chen X, Abdul-Ghani M, Cersosimo E, Del Prato S, DeFronzo R. Increase in Endogenous Glucose Production With SGLT2 Inhibition Is Unchanged by Renal Denervation and Correlates Strongly With the Increase in Urinary Glucose Excretion. Diabetes Care. 2020 May;43(5):1065-1069. doi: 10.2337/dc19-2177. Epub 2020 Mar 6. PMID 32144165

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Diabetic and non-diabetic subjects were assigned to both interventions after randomization, either dapagliflozin first with placebo second, or placebo first and then dapagliflozin next.
Groups:
- Dapagliflozin First - Diabetic: Subjects who have undergone renal transplant are randomly assigned to receive either dapagliflozin first followed by the placebo
- Placebo Oral Tablet First - Diabetic: Subjects who have undergone renal transplant are randomly assigned to receive placebo first followed by dapagliflozin
- Dapagliflozin First - Non-diabetic: Non-diabetic subjects who have undergone renal transplant are randomly assigned to dapagliflozin first and then receive placebo
- Placebo Oral Tablet First - Non-diabetic: Non-diabetic subjects who have undergone renal transplant are randomly assigned to placebo first and then receive dapagliflozin
- Control Group: Type 2 Diabetic subjects who did not undergo renal transplant and received dapagliflozin
Period: Overall Study
Arm/Group | Dapagliflozin First - Diabetic | Placebo Oral Tablet First - Diabetic | Dapagliflozin First - Non-diabetic | Placebo Oral Tablet First - Non-diabetic | Control Group
Started | 3 | 3 | 4 | 4 | 20
Completed | 3 | 3 | 4 | 4 | 20
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects who underwent renal transplant surgery with intact native kidneys, and a type 2 diabetic control group that did not undergo renal transplant
Groups:
- Diabetic Subjects: Diabetic renal transplant subjects with native kidneys intact who were Type 2 diabetics
- Non-diabetic Subjects: Non-diabetic subjects after renal transplant with intact native kidneys
- Control Group: Type 2 diabetic subjects who did not under go renal transplant
- Total: Total of all reporting groups
Arm/Group | Diabetic Subjects | Non-diabetic Subjects | Control Group | Total
Number analyzed (Participants) | 6 | 8 | 20 | 34
Age, Customized [Count of Participants; unit: Participants]
  Subjects between 18 and 70 years | 6 | 8 | 20 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 8 | 17
  Male | 0 | 5 | 12 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 6 of the subjects analyzed were diabetic and the remaining 8 were non-diabetic
  Participants
    Hispanic | 5 | 5 | 12 | 22
    White Non-Hispanic | 1 | 1 | 8 | 10
    Black Non-Hispanic | 0 | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 20 | 34
A1C (average blood glucose level over 3 months) [Mean (Standard Deviation); unit: Percentage of glycated hemoglobin] | 7.2 (0.1) | 5.6 (0.1) | 7.5 (0.2) | 6.4 (0.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Endogenous Glucose Production (EGP)
Description: Renal transplant subjects with native kidneys intact underwent measurement of EGP with an 8 hour infusion of 3-3H-glucose on 2 separate days with the administration in random order of either dapagliflozin 10mg or placebo after 3 hours of the tracer equilibration period. The equilibration at 3 hours was considered the baseline measurement. Measurement of change in endogenous glucose production was obtained for all subjects.
Time Frame: baseline and 240-300 minutes
Population: The control group did not have renal surgery and were only administered the dapagliflozin, not the placebo, so no participants show for baseline or 240 to 300 minutes for placebo measurements, only for dapagliflozin.
Measure: Mean (Standard Deviation); unit: mg/kg.min
Groups:
- Diabetic Subjects: Renal transplant subjects with native kidneys intact who were Type 2 diabetics
- Control Group: Type 2 diabetic subjects who did not undergo renal surgery and received dapagliflozin
Arm/Group | Diabetic Subjects | Non-diabetic Subjects | Control Group
Number analyzed (Participants) | 6 | 8 | 20
mg/kg.min
  Baseline Measurement Placebo: number analyzed (Participants) | 6 | 8 | 0
  Baseline Measurement Placebo | 2.03 (0.20) | 1.92 (0.10) |
  240-300 minute measurement Placebo: number analyzed (Participants) | 6 | 8 | 0
  240-300 minute measurement Placebo | 1.55 (0.09) | 1.68 (0.10) |
  Baseline Measurement Dapagliflozin | 2.21 (0.19) | 1.85 (0.10) | 2.5 (0.1)
  240-300 minute measurement Dapagliflozin | 1.96 (0.14) | 1.78 (0.10) | 2.6 (0.1)

2. Secondary Outcome: Change in Fasting Plasma Glucose
Description: Change in Fasting Plasma Glucose in Type 2 Diabetes Mellitus subjects only
Time Frame: baseline and 240-300 minutes
Population: Only type 2 diabetic subjects were included in this group, so the 8 non-diabetic renal transplant subjects were not included.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Control Group: Subjects who are type 2 diabetics who did not undergo renal transplant
Arm/Group | Diabetic Subjects | Control Group
Number analyzed (Participants) | 6 | 20
mg/dL
  Baseline Measurement Placebo: number analyzed (Participants) | 6 | 0
  Baseline Measurement Placebo | 143 (14) |
  240-300 minute measurement Placebo: number analyzed (Participants) | 6 | 0
  240-300 minute measurement Placebo | 124 (10) |
  Baseline Measurement Dapagliflozin | 143 (15) | 135.7 (2.6)
  240-300 minute measurement Dapagliflozin | 112 (9) | 106.6 (1.3)

3. Secondary Outcome: Change in Fasting Plasma Insulin
Description: Change in Fasting Plasma Insulin in Type 2 Diabetes Mellitus subjects in diabetic subjects only
Time Frame: baseline and 240-300 minutes
Population: Only type 2 diabetic subjects were included in this group, so the 8 subjects who were non-diabetic who had renal transplant were not included.
Measure: Mean (Standard Deviation); unit: U/ml
Arm/Group | Diabetic Subjects | Control Group
Number analyzed (Participants) | 6 | 20
U/ml
  Baseline Measurement Placebo: number analyzed (Participants) | 6 | 0
  Baseline Measurement Placebo | 12 (2) |
  240-300 minute measurement Placebo: number analyzed (Participants) | 6 | 0
  240-300 minute measurement Placebo | 10 (1.1) |
  Baseline Measurement Dapagliflozin | 14 (3) | 15.2 (1.9)
  240-300 minute measurement Dapagliflozin | 11 (2) | 9.9 (1.2)

ADVERSE EVENTS:
Time Frame: Baseline to 8 hours
Groups:
- Diabetic Subjects Dapagliflozin: Diabetic subjects who have undergone kidney surgery, and have a dapagliflozin infusion
- Diabetic Subjects Placebo: Diabetic subjects who have undergone kidney surgery, and have a placebo infusion
- Non-diabetic Subjects Dapagliflozin: Non-Diabetic subjects who have undergone kidney surgery, and have a dapagliflozin infusion
- Non-diabetic Subjects Placebo: Non-Diabetic subjects who have undergone kidney surgery, and have a placebo infusion
- Control Group: Type 2 Diabetic subjects who have not undergone renal surgery
Arm/Group | Diabetic Subjects Dapagliflozin | Diabetic Subjects Placebo | Non-diabetic Subjects Dapagliflozin | Non-diabetic Subjects Placebo | Control Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/8 | 0/8 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/8 | 0/8 | 0/20
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/8 | 0/8 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/95/NCT03168295/Prot_SAP_000.pdf